CLINICAL TRIAL: NCT01329198
Title: Scheduled and Responsive Brain Stimulation for the Treatment of Tourette Syndrome
Brief Title: Brain Stimulation for the Treatment of Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 414-2008- A
Record Dates: First submitted 2011-03-25; First posted 2011-04-05 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Tourette Syndrome
Keywords: tourette; tourette's; TS; tourette syndrome; tourette's syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective blinded staggered onset design
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Programming to be performed for this study by the programming investigator under the supervision of the PI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Delayed Activation - Deep Brain Stimulation (DBS) (Active Comparator): Delayed Activation stimulation in which no electrical charge is delivered through the Neuropace RNS (responsive neurostimulation) system for the first 59 days. On Day 60, all subjects will be programmed to receive active stimulation.
  * There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (3 subjects in each group) will undergo identical programming procedures at 30 and 60 days.
  Interventions: Device: NeuroPace RNS® System Deep Brain Stimulator
- Immediate Activation - Deep Brain Stimulation (DBS) (Active Comparator): Active stimulation through the Neuropace RNS (responsive neurostimulation) system at settings to maximally reduce tic frequency & severity, while limiting potential stimulation-induced side-effects.
  * There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (3 subjects in each group) will undergo identical programming procedures at 30 and 60 days.
  Interventions: Device: NeuroPace RNS® System Deep Brain Stimulator

INTERVENTIONS:
Device: NeuroPace RNS® System Deep Brain Stimulator — Utilizes a signal that the device detects and will respond to with an electrical pre-defined pulse if the signal is encountered.
  Other Names: NeuroPace DBS (deep brain stimulation)

SUMMARY:
The purpose of this trial is to determine whether a particular type of Deep Brain Stimulation (DBS), scheduled Deep Brain stimulation (SBS), is an effective and safe treatment for Tourettte syndrome (TS).

The trial will also examine the brain activity associated with TS and tics and explore the possibility of responsive brain stimulation (RBS).

DETAILED DESCRIPTION:
DBS is a surgical procedure that seeks to change the brain's electrical signalling by means of applied electrical current. To this end, a wire with tiny stimulating electrodes is implanted into one or both sides of the brain. An electrode is a small piece of metal used to take an electric current to or from a power source. These electrodes are connected under the skin on the scalp to a small electrical unit called an INS (implantable neurostimulator), which is similar to a heart pacemaker. The device sends out electrical impulses that appear to change the normal flow of electricity in the brain.

The wires which house the electrodes will be implanted on both sides of the brain oriented towards the centromedian thalamus-parafascicular complex. This region of the brain has to date the greats number of documented cases revealing significant improvements in motor tics.

This region of the brain will also provide a target where physiological changes related to motor tics are likely to be discovered.

The device we propose for this study has several features that make it more suitable for use in the TS population than other devices. It is self-contained in the skull and brain, and contains no tunneled neck connector wire and no chest pacemaker deice. This will help to lessen infection, and will assist in limiting device-related fractures due to tics involving neck region. Also, the system can record electro-encephalograph data from the area of the electrodes, which will assist us in gathering information about what specific physiological changes are correlated with tics.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of TS must be made by both a neurologist and a psychiatrist and must meet standardized criteria
* must have a minimum score on the primary tic rating scale
* symptoms must be causing significant impairment in functioning, making it impossible or almost impossible to do daily activities, including work or school and interactions with friends and family, causing severe distress and a poor quality of life
* symptoms have not responded well enough to medications prescribed by a neurologist or psychiatrist experienced in treating TS. Must have had trials of drugs from three different classes of drugs that have not worked.
* must have received stable and effective treatment of any other existing medical or psychological problems for the past 6 months.
* current TS related-medication(s) must be stable for at least a month without a dose change prior to surgery and must be willing to keep these medications stable and unchanged throughout the study or must be off of TS-related medications for at least three months prior to surgery
* If tics involve only one group of muscles or might be controllable by botulinum toxin treatment, must try botulinum treatment before considering surgery.
* must have a negative urine drug screen
* must give informed consent

Exclusion Criteria:

* have a simple motor tic or movement disorder other than TS, or medication-related movement disorders from TS medications
* have had any previous brain surgery including deep brain stimulation, ablative capsulotomy or cingulotomy
* have another psychiatric condition (including body dysmorphic disorder, a delusional disorder or a biological brain disorder), dementia or cognitive dysfunction that would place subject at risk for worsening cognition and/or may impact ability to comply with study procedures. Also included is any other psychiatric disorder that requires medications or treatments that would interfere with the functioning of the DBS device.
* have any significant substance abuse or dependence (e.g., stimulants, alcohol, opiates, benzodiazepines) within the past six months
* have a severe medical disease including cardiovascular disorder, lung disorder, kidney disease, chronic neurological disease, hematological disease, or frailty that impacts tolerability of the surgery as judged by the screening physicians
* pre-surgery MRI is considered abnormal. You may also be excluded if your brain is considered very small.
* have a history of serious suicidal behavior, are unable to control suicide attempts, or are currently at risk of suicide, in the judgement of the investigator
* have head-banging tics or tics that have the potential to damage the RNS System
* are currently pregnant or breast-feeding, plan to become pregnant during the study, or are not using effective contraception
* are currently enrolled in another investigational study
* have an implant such as a pacemaker or neurostimulator containing electrical circuitry or that generates electrical signals
* have any metal orthopedic pins or plates, metal orthodontics, or non-removable body jewelry
* require diathermy treatments during physical or occupational therapy
* have a problem that will require repeat Magnetic Resonance Imaging (MRI) scans

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Okun, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Movement Disorders Center, Gainesville, Florida, United States

REFERENCES:
- [Derived] Okun MS, Foote KD, Wu SS, Ward HE, Bowers D, Rodriguez RL, Malaty IA, Goodman WK, Gilbert DM, Walker HC, Mink JW, Merritt S, Morishita T, Sanchez JC. A trial of scheduled deep brain stimulation for Tourette syndrome: moving away from continuous deep brain stimulation paradigms. JAMA Neurol. 2013 Jan;70(1):85-94. doi: 10.1001/jamaneurol.2013.580. PMID 23044532
- See also: Increased Thalamic Gamma Band Activity Correlates with Symptom Relief following Deep Brain Stimulation in Humans with Tourette's Syndrome — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3435399/

RESULTS

PARTICIPANT FLOW:
Groups:
- Delayed Activation DBS: Sham stimulation in which no electrical charge is delivered through the Neuropace RNS system. By Day 60, all subjects will be programmed to receive active stimulation.
  * There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (will undergo identical programming procedures at 30 and 60 days.
- Immediate Activation DBS: Active stimulation through the Neuropace RNS system at settings to maximally reduce tic frequency & severity, while limiting potential stimulation-induced side-effects
  * There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (3 subjects in each group) will undergo identical programming procedures at 30 and 60 days.
Period: Overall Study
Arm/Group | Delayed Activation DBS | Immediate Activation DBS
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Delayed Activation DBS: Sham stimulation in which no electrical charge is delivered through the Neuropace RNS system. By Day 60, all subjects will be programmed to receive active stimulation.
  * There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (3 subjects in each group) will undergo identical programming procedures at 30 and 60 days.
- Total: Total of all reporting groups
Arm/Group | Delayed Activation DBS | Immediate Activation DBS | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Yale Global Tic Severity Scale (YGTSS) Scores From Baseline to 6 Months Across All Study Participants Presented
Description: The Yale Global Tic Severity Scale (YGTSS) is a semistructured clinician-rated instrument that assesses the severity and frequency of motor and phonic tics over the previous week. Five index scores are obtained during the assessment, where higher scores indicate greater frequency or severity. These indices are:
  * Total Motor Tic Score (0-25)
  * Total Phonic Tic Score (0-25
  * Total Tic Score (0-50)
  * Overall Impairment Rating (0-50)
  * Global Severity Score (0-7)
  The YGTSS Total Score is obtained by adding the Total Tic Score to the Overall Impairment Rating. The efficacy of the intervention will be assessed by comparing each subject's 6-month YGTSS Total Score to the pre-operative value for the same patient. Efficacy is considered 50% or greater reduction in this score.
Time Frame: Baseline to 6 Months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Delayed Activation DBS | Immediate Activation DBS
Number analyzed (Participants) | 3 | 2
units on a scale
  Change in YGTSS Baseline to 6 months | -20.33 [-41.46 to 0.79] | -14.05 [-127.77 to 99.67]
  YGTSS Baseline Score | 91 [79.47 to 102.53] | 92.5 [86.14 to 98.86]
  YGTSS 6 Month Score | 70.67 [63.65 to 77.69] | 78.45 [59.43 to 97.47]
Statistical Analysis 1: Comparison: Delayed Activation DBS vs Immediate Activation DBS; Test type: Superiority; p = 0.013, ANOVA; Mean Difference (Final Values) = -17.8, Standard Deviation 9.4 — Mean change in YGTSS scores from Baseline to 6 Months across all study participants presented

2. Secondary Outcome: Correlation of Tics and Neural Physiology
Description: Electrical recordings of electroencephalography activity were taken from each subject's implanted leads at each visit from baseline to 6 months. At baseline, the recordings were taken with the device in the off state (not stimulating), while at the 6 month visits the recordings were taken with the subject's device set to optimal parameters for tic control. Using Pearson's correlation coefficient, the variations in frequency and power which were observed were correlated with the Yale Global Tic Severity (YGTSS) scores obtained during primary outcome testing.
Time Frame: Baseline to 6 Months
Measure: Number; unit: Pearson Correlation Coefficient
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4 | Subject 5
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1
Pearson Correlation Coefficient | -0.317 | -0.950 | -0.704 | -0.855 | -0.399

ADVERSE EVENTS:
Time Frame: Adverse event data was collected starting the day of the screening visit and continuing through each subject's 2 year follow-up visit.
Groups:
- Sham DBS: Sham stimulation in which no electrical charge is delivered through the Neuropace RNS system.
  NeuroPace RNS® System Deep Brain Stimulator: • There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (3 subjects in each group) will undergo identical programming procedures at 30 and 60 days.
- Active DBS: Active stimulation through the Neuropace RNS system at settings to maximally reduce tic frequency & severity, while limiting potential stimulation-induced side-effects
  NeuroPace RNS® System Deep Brain Stimulator: • There will be a one month post-operative period during which stimulation is not turned on.
  * One month post-implant, subjects will be randomized one to one in a blinded fashion to receive active or sham stimulation.
  * By Day 60, all subjects will be programmed to receive active stimulation. Physiological data will be collected for Specific Aim 2 of the study.
  * Both the sham and the active groups (3 subjects in each group) will undergo identical programming procedures at 30 and 60 days.
Arm/Group | Sham DBS | Active DBS
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham DBS (N=3) | Active DBS (N=2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Attempted suicide (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sham DBS (N=3) | Active DBS (N=2)
Paresthesia (Nervous system disorders) | 3 (25) | 2 (18) — During stimulation testing, varying configurations of settings would induce different sensations - tingling, numbness, pressure, cold and warmth.
Presyncope (Nervous system disorders) | 3 (10) | 2 (4) — Stimulation-induced feelings of dizziness or lightheadedness
Movements Involuntary (Nervous system disorders) | 3 (7) | 2 (2) — Stimulation-induced pulling of the head or neck to one side or another.
Dysarthria (Nervous system disorders) | 1 (1) | 1 (2) — During stimulation testing, a sudden inability to form words.
Blurred vision (Eye disorders) | 3 (5) | 2 (5)
Nausea (Gastrointestinal disorders) | 2 (4) | 1 (1) — Stimulation-induced abdominal uneasiness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No